CLINICAL TRIAL: NCT04396028
Title: Assessment of the Pulmonary Area in Newborn With Congenital Diaphragmatic Hernia: a Retrospective Analysis of Respiratory Function, Risk of Recurrence and Mortality
Brief Title: Measurement of Lung Area at Chest Radiography to Define the Prognosis in Newborns With CDH
Acronym: NeoAPACHE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Giacomo Cavallaro, Principal Investigator, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Other Study IDs: OSMAMI-04/05/2020-0015998-U
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Congenital Diaphragmatic Hernia
Keywords: congenital diaphragmatic hernia; radiographic pulmonary area; lung hypoplasia; respiratory function; mortality; recurrence
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital; Respiratory Aspiration; Recurrence | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: data collection — retrospective data collection

SUMMARY:
CDH represents a malformative disorder characterized by an incomplete diaphragm formation. This results in poor lung development (pulmonary hypoplasia), associated with altered vascularization of the lung (pulmonary hypertension), determining respiratory and cardiovascular insufficiency at birth. CDH shows high mortality and significant morbidity so that its prognostic evaluation remains challenging.

The measurement of lung area at chest radiography is considered an alternative method to assess lung development in the newborn. A correlation between lung area and functional residual capacity (FRC) was demonstrated in newborns with CDH.

However, the relationship between lung area and other aspects of respiratory function has never been investigated. Since CDH compromises lung development as a whole, it is likely to assume that lung area at birth may have an impact on patient's performance at pulmonary function tests during follow-up. In particular, as lung area increased, a trend towards normalization in respiratory function would be expected.

Moreover, the role of the radiographic area at birth as a possible predictor of death should be further characterized, aiming to clarify the complex association between lung area and mortality, which is strongly influenced by both pulmonary hypoplasia and pulmonary hypertension.

The principal aim of this study is to determine if changes in the radiographic pulmonary area measured on the first day of life are related to patients' pulmonary function at one year of life, considering two main respiratory parameters: tidal volume (VT) and respiratory rate (RR).

Secondary objectives are the analysis of the association between radiographic pulmonary area and: 1) risk of death during the first year of life; 2) risk of hernia recurrence during the first year of life.

The investigators will retrospectively consider a cohort of newborns with CDH. For each patient, the investigators will measure lung area at chest radiography performed preoperatively within 24 hours after birth and will collect data regarding demographics, clinical course, and follow-up.

Through our study, the investigators aim to improve the current understanding of the role of radiographic lung area in characterizing lung development and prognosis in CDH patients. The investigators believe that this could become a low-cost and straightforward tool that will assist the clinician in making decisions regarding the patient's management and follow up.

DETAILED DESCRIPTION:
The study period considered will be January 2012 - December 2018. From the medical record of each patient, the investigators will collect the following data: prenatal history, hernia severity, fetal endoscopic tracheal occlusion (FETO) procedure, demographics, respiratory insufficiency, and mechanical ventilation, cardiocirculatory insufficiency and pharmacological hemodynamic support, pulmonary hypertension and need for pulmonary vasodilators, need for extracorporeal life support (ECMO), comorbidities, timing of surgical repair, use of prosthetic patch, intra- and post-operative complications, clinical and instrumental follow-up, pulmonary function tests, recurrence, death. The confidentiality of all data will be maintained.

Regarding the assessment of the radiographic pulmonary area, two operators (a neonatologist and a pediatric radiologist) will independently review all preoperative digital radiograms performed within 24 hours of life. For each patient, the radiogram showing the best lung-recruitment will be selected. Lung area will be assessed by freehand tracing of the perimeter of the thoracic area, as outlined by the diaphragm and the rib cage, excluding the mediastinal structures and abdominal contents herniated in the thorax. The only aerated portion of the lungs will be considered. The corresponding area will be automatically calculated by the software. Three measures will be performed: 1) ipsilateral lung area (cm2); 2) contralateral lung area (cm2); 3) total lung area (cm2), derived from the sum of the preceding two. The agreement between lung measurements performed by the two operators will be evaluated to verify the reproducibility of the method.

Pulmonary function test performed during spontaneous sleeping at the age of 1 year will be reviewed. The measurements of VT and RR will be recorded. The predicted value of VT and RR will be obtained, and their Z-Score will be calculated using reference equations of a population of healthy children. Z-Score is a numerical measure used to express how much an observed value deviates from the mean expected normal value in terms of standard deviation.

ELIGIBILITY:
Inclusion Criteria:

* Inborn and outborn patients admitted to the NICU within 24 hours after birth.
* Prenatal or postnatal (within 24 hours after birth) diagnosis of CDH.
* Preoperative chest radiograph performed for clinical purposes within 24 hours after birth in our NICU.

Exclusion Criteria:

* Diagnosis of CDH made beyond 24 hours after birth
* Admission to the NICU beyond 24 hours after birth
* Preoperative chest radiograph performed beyond 24 hours after birth, rotated/asymmetric, with air leak (pneumothorax, pneumoperitoneum), not performed in our NICU or not accessible
* Early death (within 1 hour after birth)

Ages: 1 Hour to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants with CDH born between January 2012 and December 2018, hospitalized at birth or within 24 hours of life at the Neonatal Intensive Care Unit of Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy, and followed-up longitudinally during the first year of life.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2020-07-09 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Association between radiographic pulmonary area and respiratory function | 12 months
  To evaluate the association between changes in radiographic pulmonary area at birth and trend in VT and RR measured at pulmonary function tests performed during follow-up at the age of 1 year. The association will be studied through linear regression models.

SECONDARY OUTCOMES:
Association between radiographic pulmonary area and mortality | 12 months
  To evaluate the association between changes in radiographic pulmonary area and the risk of death during the first year of life, following logistic regression models.
Association between radiographic pulmonary area and hernia recurrence | 12 months
  To evaluate the association between changes in radiographic pulmonary area and the risk of hernia recurrence during the first year of life, following logistic regression models.

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Cavallaro, MD, PhD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Neonatal Intensive Care Unit, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan, MI, Italy

REFERENCES:
- [Background] Deprest J, Brady P, Nicolaides K, Benachi A, Berg C, Vermeesch J, Gardener G, Gratacos E. Prenatal management of the fetus with isolated congenital diaphragmatic hernia in the era of the TOTAL trial. Semin Fetal Neonatal Med. 2014 Dec;19(6):338-48. doi: 10.1016/j.siny.2014.09.006. Epub 2014 Nov 11. PMID 25447987
- [Background] Snoek KG, Greenough A, van Rosmalen J, Capolupo I, Schaible T, Ali K, Wijnen RM, Tibboel D. Congenital Diaphragmatic Hernia: 10-Year Evaluation of Survival, Extracorporeal Membrane Oxygenation, and Foetoscopic Endotracheal Occlusion in Four High-Volume Centres. Neonatology. 2018;113(1):63-68. doi: 10.1159/000480451. Epub 2017 Oct 28. PMID 29080897
- [Background] Coughlin MA, Werner NL, Gajarski R, Gadepalli S, Hirschl R, Barks J, Treadwell MC, Ladino-Torres M, Kreutzman J, Mychaliska GB. Prenatally diagnosed severe CDH: mortality and morbidity remain high. J Pediatr Surg. 2016 Jul;51(7):1091-5. doi: 10.1016/j.jpedsurg.2015.10.082. Epub 2015 Nov 10. PMID 26655216
- [Background] Bagolan P, Morini F. Long-term follow up of infants with congenital diaphragmatic hernia. Semin Pediatr Surg. 2007 May;16(2):134-44. doi: 10.1053/j.sempedsurg.2007.01.009. PMID 17462566
- [Background] American Academy of Pediatrics Section on Surgery; American Academy of Pediatrics Committee on Fetus and Newborn; Lally KP, Engle W. Postdischarge follow-up of infants with congenital diaphragmatic hernia. Pediatrics. 2008 Mar;121(3):627-32. doi: 10.1542/peds.2007-3282. PMID 18310215
- [Background] Rocha G, Azevedo I, Pinto JC, Guimaraes H. Follow-up of the survivors of congenital diaphragmatic hernia. Early Hum Dev. 2012 Apr;88(4):255-8. doi: 10.1016/j.earlhumdev.2011.08.025. Epub 2011 Sep 23. PMID 21945360
- [Background] Chen C, Jeruss S, Chapman JS, Terrin N, Tighiouart H, Glassman E, Wilson JM, Parsons SK. Long-term functional impact of congenital diaphragmatic hernia repair on children. J Pediatr Surg. 2007 Apr;42(4):657-65. doi: 10.1016/j.jpedsurg.2006.12.013. PMID 17448762
- [Background] Jancelewicz T, Chiang M, Oliveira C, Chiu PP. Late surgical outcomes among congenital diaphragmatic hernia (CDH) patients: why long-term follow-up with surgeons is recommended. J Pediatr Surg. 2013 May;48(5):935-41. doi: 10.1016/j.jpedsurg.2013.02.005. PMID 23701763
- [Background] Dimitriou G, Greenough A, Kavvadia V, Shute M, Karani J. A radiographic method for assessing lung area in neonates. Br J Radiol. 1999 Apr;72(856):335-8. doi: 10.1259/bjr.72.856.10474492.
- [Background] May C, Prendergast M, Salman S, Rafferty GF, Greenough A. Chest radiograph thoracic areas and lung volumes in infants developing bronchopulmonary dysplasia. Pediatr Pulmonol. 2009 Jan;44(1):80-5. doi: 10.1002/ppul.20952. PMID 19085927
- [Background] Dassios T, Curley A, Krokidis M, Morley C, Ross-Russell R. Correlation of radiographic thoracic area and oxygenation impairment in bronchopulmonary dysplasia. Respir Physiol Neurobiol. 2016 Jan;220:40-5. doi: 10.1016/j.resp.2015.09.009. Epub 2015 Sep 26. PMID 26410458
- [Background] Dimitriou G, Greenough A, Davenport M, Nicolaides K. Prediction of outcome by computer-assisted analysis of lung area on the chest radiograph of infants with congenital diaphragmatic hernia. J Pediatr Surg. 2000 Mar;35(3):489-93. doi: 10.1016/s0022-3468(00)90219-7. PMID 10726694
- [Background] Dassios T, Ali K, Makin E, Bhat R, Krokidis M, Greenough A. Prediction of Mortality in Newborn Infants With Severe Congenital Diaphragmatic Hernia Using the Chest Radiographic Thoracic Area. Pediatr Crit Care Med. 2019 Jun;20(6):534-539. doi: 10.1097/PCC.0000000000001912. PMID 30925570
- [Background] Putnam LR, Gupta V, Tsao K, Davis CF, Lally PA, Lally KP, Harting MT; Congenital Diaphragmatic Hernia Study Group. Factors associated with early recurrence after congenital diaphragmatic hernia repair. J Pediatr Surg. 2017 Jun;52(6):928-932. doi: 10.1016/j.jpedsurg.2017.03.011. Epub 2017 Mar 16. PMID 28359590
- [Background] Al-Iede MM, Karpelowsky J, Fitzgerald DA. Recurrent diaphragmatic hernia: Modifiable and non-modifiable risk factors. Pediatr Pulmonol. 2016 Apr;51(4):394-401. doi: 10.1002/ppul.23305. Epub 2015 Sep 7. PMID 26346806
- [Background] Nguyen TT, Hoo AF, Lum S, Wade A, Thia LP, Stocks J. New reference equations to improve interpretation of infant lung function. Pediatr Pulmonol. 2013 Apr;48(4):370-80. doi: 10.1002/ppul.22656. Epub 2012 Sep 4. PMID 22949414
- [Background] Van der Veeken L, Russo FM, De Catte L, Gratacos E, Benachi A, Ville Y, Nicolaides K, Berg C, Gardener G, Persico N, Bagolan P, Ryan G, Belfort MA, Deprest J. Fetoscopic endoluminal tracheal occlusion and reestablishment of fetal airways for congenital diaphragmatic hernia. Gynecol Surg. 2018;15(1):9. doi: 10.1186/s10397-018-1041-9. Epub 2018 May 8. PMID 29770109
- [Background] Snoek KG, Reiss IK, Greenough A, Capolupo I, Urlesberger B, Wessel L, Storme L, Deprest J, Schaible T, van Heijst A, Tibboel D; CDH EURO Consortium. Standardized Postnatal Management of Infants with Congenital Diaphragmatic Hernia in Europe: The CDH EURO Consortium Consensus - 2015 Update. Neonatology. 2016;110(1):66-74. doi: 10.1159/000444210. Epub 2016 Apr 15. PMID 27077664
- [Background] Hollinger LE, Buchmiller TL. Long term follow-up in congenital diaphragmatic hernia. Semin Perinatol. 2020 Feb;44(1):151171. doi: 10.1053/j.semperi.2019.07.010. Epub 2019 Jul 31. PMID 31451197
- [Derived] Amodeo I, Pesenti N, Raffaeli G, Macchini F, Condo V, Borzani I, Persico N, Fabietti I, Bischetti G, Colli AM, Ghirardello S, Gangi S, Colnaghi M, Mosca F, Cavallaro G. NeoAPACHE II. Relationship Between Radiographic Pulmonary Area and Pulmonary Hypertension, Mortality, and Hernia Recurrence in Newborns With CDH. Front Pediatr. 2021 Jul 12;9:692210. doi: 10.3389/fped.2021.692210. eCollection 2021. PMID 34322463
- [Derived] Amodeo I, Borzani I, Corsani G, Pesenti N, Raffaeli G, Macchini F, Condo V, Persico N, Ghirardello S, Colnaghi M, Mosca F, Cavallaro G. Fetal MRI mediastinal shift angle and respiratory and cardiovascular pharmacological support in newborns with congenital diaphragmatic hernia. Eur J Pediatr. 2022 Jan;181(1):323-334. doi: 10.1007/s00431-021-04207-8. Epub 2021 Jul 23. PMID 34302257
- [Derived] Amodeo I, Raffaeli G, Pesenti N, Macchini F, Condo V, Borzani I, Persico N, Fabietti I, Ophorst M, Ghirardello S, Gangi S, Colnaghi M, Mosca F, Cavallaro G. The NeoAPACHE Study Protocol I: Assessment of the Radiographic Pulmonary Area and Long-Term Respiratory Function in Newborns With Congenital Diaphragmatic Hernia. Front Pediatr. 2020 Oct 30;8:581809. doi: 10.3389/fped.2020.581809. eCollection 2020. PMID 33194913